CLINICAL TRIAL: NCT01560494
Title: Validation of a Structured Training and Assessment Curriculum (STAC) for Technical Skill Acquisition in Minimally Invasive Surgery. A Randomized Controlled Study
Brief Title: Validation of a Curriculum (STAC) for Technical Skill Acquisition in Minimally Invasive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: STAC
Record Dates: First submitted 2012-03-13; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Surgical Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- STAC curriculum (Experimental)
  Interventions: Other: STAC curriculum
- Conventional Curriculum (No Intervention)

INTERVENTIONS:
Other: STAC curriculum — The STAC curriculum consists of theoretical preparation, case-based learning, proficiency-based virtual reality training, laparoscopic box training, and operating room participation.
  Arms: STAC curriculum

SUMMARY:
This study describes the development and validation of a structured training and assessment curriculum (STAC) for a basic laparoscopic procedure. The investigators hypothesized that residents trained using the STAC curriculum would demonstrate superior technical skills in the operating room compared to residents that were trained using a traditional curriculum.

DETAILED DESCRIPTION:
The objective of this study was to develop and validate an ex-vivo comprehensive curriculum for a basic laparoscopic procedure. Although simulators have been well validated as tools to teach technical skills, their integration into comprehensive curricula is lacking. Moreover, neither the effect of ex-vivo training on learning curves in the operating room (OR), nor the effect on non-technical proficiency has been investigated. This randomized single-blinded prospective trial allocated 20 surgical trainees to a structured-curriculum (STAC) group or conventional residency training. The STAC curriculum consisted of: case-based learning, proficiency-based virtual reality training, laparoscopic box training, and OR participation. After completion of the intervention, all participants performed 5 sequential laparoscopic cholecystectomies in the OR. The primary outcome measure was the difference in technical performance between the 2 groups during the first laparoscopic cholecystectomy. Secondary outcome measures included differences with respect to: learning curves in the OR, technical proficiency of each sequential laparoscopic cholecystectomy, and non-technical skills.

ELIGIBILITY:
Inclusion Criteria:

* post graduate year 1 and 2 general surgical residents
* completed less than 10 laparoscopic cholecystectomies or appendectomies as the primary surgeon

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Technical skills | 6 months
  Participants' technical skills will be assessed in the operating room as they perform a laparoscopic cholecystectomy under supervision. The procedure will be video-recorded and sent for assessment to a blinded evaluator. Technical skills will be assessed using a previously validated technical skills assessment tool (Objective Structured Assessment of Technical Skill - OSATS)

SECONDARY OUTCOMES:
cognitive knowledge | 6 months
  Study participants will complete a multiple choice quiz designed to assess congitive knowledge relating to performing laparoscpoic cholecystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Teodor Grantcharov, MD, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Palter VN, Orzech N, Reznick RK, Grantcharov TP. Validation of a structured training and assessment curriculum for technical skill acquisition in minimally invasive surgery: a randomized controlled trial. Ann Surg. 2013 Feb;257(2):224-30. doi: 10.1097/SLA.0b013e31827051cd. PMID 23013806